CLINICAL TRIAL: NCT03175705
Title: A Study of Specific HCC Antigens CD8+ T Cells Therapy for Treating Patients With Relapsed/Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Adoptive Transfer of Specific HCC Antigens CD8+ T Cells for Treating Patients With Relapsed/Advanced HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, LU JUN, Director of Hepatology and Cancer Biotherapy Ward, Beijing YouAn Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beijing Youan Ethics[2017]06
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interleukin-2; Tegafur; gimeracil; potassium oxonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous T cell therapy+Tegafur+Interleukin-2 (IL-2) (Experimental): Autologous in vitro expanded HCC antigens-specific CD8+ T lymphocytes in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with relapsed/advanced HCC.
  Interventions: Biological: HCC antigens-specific CD8+ T lymphocytes; Drug: IL-2; Drug: Tegafur

INTERVENTIONS:
Biological: HCC antigens-specific CD8+ T lymphocytes — Three different dosing schedules will be evaluated. Three patients will be evaluated on each dosing schedule.
  The following dose levels will be evaluated:
  Loading Dose 1: 3x10^7/m2 Loading Dose 2: 6x10^7/m2 Loading Dose 3: 9x10^7/m2 The doses are calculated according to the actual number of GPC3/NY-ESO-1/AFP specific cytotoxic lymphocytes (CTLs)
Drug: IL-2 — IL-2 will be given at a dose of 25000 IU/kg/day for 5-14 days.
  Other Names: Human recombinated Interleukin-2
Drug: Tegafur — Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Other Names: Gimeracil and Oteracil potassium Capsules

SUMMARY:
This study enrolls patients who have relapsed/advanced hepatocellular carcinoma (HCC, BCLC stage C). The HCC tumor relapsed or metastasized through the body after standard treatment or the patients cannot receive standard treatment under current conditions. This research study uses specific HCC antigens CD8+ T cells, a new experimental treatment.

The purpose of this study is to evaluate the safety and tolerance as well as the potential clinical efficacy of an adoptive transfer of CD8+ T cells, sorted with human leukocyte antigen (HLA)-peptide multimers and specific for Glypican (GPC)-3 /New York Esophageal Squamous-1 (NY-ESO-1) /alpha-fetoprotein (AFP) antigens and cultured in vitro, to patients suffering from relapsed/advanced hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Patients with relapsed/advanced HCC (BCLC, stage C) proved by histopathology or proved by CT or MRI imaging system, proven GPC3/NY-ESO-1/AFP(+), relapsed after previous therapy and no effective therapies known at this time.
* Life expectancy of ≥ 12 weeks.
* WBC>3.5×10^9/L, LYMPH> 0.8×10^9/L, Hb>85g/L, PLT>50×10^9/L, Cre<1.5×the upper limit of normal value.
* Able to understand and sign the informed consent.

Exclusion Criteria:

* Any uncontrolled systematic disease: hypertension, heart disease, and et al.;
* Portal vein tumor thrombus, central nervous system tumor metastasis, or combined with other tumors;
* Receiving radiochemotherapy, local therapy, or targeting drugs within 4 weeks prior to this treatment;
* Unstable immune systematic diseases or Infectious diseases;
* Combined with AIDS or syphilis;
* Patients with history of stem cell or organ transplantation;
* Patients with allergic history to related drugs and immunotherapy;
* Patients with complications associated with liver diseases: moderate or severe pleural effusion, pericardial effusion, ascites, or gastrointestinal hemorrhage;
* Pregnant or lactating subjects;
* Unsuitable subjects considered by clinicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 4 weeks
  Defined as signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

SECONDARY OUTCOMES:
Biological activity of infused T cells | 4 weeks
  To assess the biological activity of infused in vitro expanded and sorted HCC antigens-specific T cells.

OTHER OUTCOMES:
Progress Free Survival (PFS) | 12 weeks or up to death
  PFS is the time that passes from the date that patient enrolled in the clinical trial and the date on which HCC progresses or the date on which the patient dies. HCC progression was evaluated by imaging according to the irRC standard.
Disease Control Rate (DCR) | 12 weeks or up to death
  DCR is the proportion of patients who had a response rate including complete remission (CR), partial remission (PR) and disease stabilization (SD) evaluated by imaging according to the irRC standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided